CLINICAL TRIAL: NCT05926414
Title: A Prospective, Multi-Center, Observational Study to Evaluate the Efficacy and Safety of Envlo Tablet or Envlomet SR Tablet in Patients With Type II Diabetes Mellitus
Brief Title: To Evaluate the Efficacy and Safety of Envlo Tablet or Envlomet SR Tablet in Patients With Type II Diabetes Mellitus
Status: Active, not recruiting | Type: Observational
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: DWENV_DB_01
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Enavogliflozin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient diagnosed with type2 diabetes mellitus: patient diagnosed with type2 diabetes mellitus
  Interventions: Drug: Enavogliflozin

INTERVENTIONS:
Drug: Enavogliflozin — treated with Envlo tab. 0.3mg
  Other Names: Envlo Tablet
Drug: Enavogliflozin — Envlomet SR Tablet 0.3/1,000mg
  Other Names: Envlomet SR Tablet

SUMMARY:
This observation study is designed as a prospective, multi-organ observation study to confirm the blood sugar control effect and safety of ENVLO tablet or Envlomet SR Tablet administration for 24 weeks in patients with type 2 diabetes who are scheduled to administer ENVLO tablet in the actual treatment environment.

DETAILED DESCRIPTION:
This observational study planned recruit population of type 2 diabetes patients who are scheduled to administer ENVLO tablet or Envlomet SR Tablet according to the medical judgment of the researcher (doctor in charge) based on permission (efficacy & effect, usage & dose, usage precautions, etc.) in the actual treatment environment.

This observational study will be conducted in an actual treatment environment regardless of whether ENVLO tablet or Envlomet SR Tablet was administered or not.

Information such as demographic information, body measurement, and vital signs performed will be collected up to 24 weeks after ENVLO tablet or Envlomet SR Tablet administration.

Data will be collected based on medical records recorded in the actual treatment environment, and there is no mandatory visit, examination, or treatment in this observation study.

ELIGIBILITY:
Inclusion Criteria:

1. an adult male and female over 19 years of age
2. A person who is a type 2 diabetic and is planed to take Envlo Tab or Envloment SR Tab for the first time according to the medical judgment of the Investigator based on the permit
3. A person who voluntarily participates in the observational study and agrees in writing to comply with the subject's precautions during the study period after hearing and understanding the detailed explanation of the characteristics of the observational study and the drug to be studied

Exclusion Criteria:

1. Persons with diabetes other than type 2 diabetes (type 1 diabetes, diabetic ketoacidosis, gestational diabetes, etc.)
2. A person who is prohibited from administering in accordance with the permission of Envlo Tab.'s

   * Patients who overreact to Envlo Tab. or Envlo Tab. components and have a history of it
   * eGFR (estimated global filtration rate) patients below 30 mL/min/1.73 m2, end-stage renal disease or on dialysis
   * Patients with moderate and severe liver failure (AST or ALT > 3x normal upper limit, Total Bilirubin > 2x normal upper limit, hepatitis or liver failure)
   * Class III or IV by classification of the New York Heart Association (NYHA)
3. Patients with unstable weight due to treatment or other treatments (surgery, diet, etc.) with obesity or weight loss medication within 3 months of Enrollment
4. Pregnant women and lactating women
5. A person who participates in another clinical trial and is administering (applying) clinical trial drugs or clinical trial medical devices
6. A person who is deemed inappropriate to participate in this observational study based on the judgment of other investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is an observational study conducted in a single group, and was calculated using the Confidence Intervals for One Mean method for the mean by referring to the average and standard deviation of changes at 12 or 24 weeks compared to the baseline of HbA1c levels in previous phase 2 and 3 clinical trials
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
change in HbA1c | at 24 weeks
  change in HbA1c at 24 weeks compared to baseline

SECONDARY OUTCOMES:
change in HbA1c | 12 weeks
  change in HbA1c at 12 weeks compared to baseline
change in FPG | 12 weeks
  change in FPG at 12 weeks compared to baseline
change in FPG | 24 weeks
  change in FPG at 24 weeks compared to baseline
percentage of subjects achieved HbA1c < 7 % | 12 weeks
  percentage of subjects achieved HbA1c < 7 % at 12 weeks compared to baseline
percentage of subjects achieved HbA1c < 7 % | 24 weeks
  percentage of subjects achieved HbA1c < 7 % at 24 weeks compared to baseline
percentage of subjects achieved HbA1c < 6.5 % | 12 weeks
  percentage of subjects achieved HbA1c < 6.5 % at 12 weeks compared to baseline
percentage of subjects achieved HbA1c < 6.5 % | 24 weeks
  percentage of subjects achieved HbA1c < 6.5 % at 24 weeks compared to baseline
therapeutic response(change in HbA1c > 0.5 % OR HbA1c < 7 %) | 12 weeks
  therapeutic response at 12 weeks compared to baseline
therapeutic response(change in HbA1c > 0.5 % OR HbA1c < 7 %) | 24 weeks
  therapeutic response at 24 weeks compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- NaRi Kim, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided